CLINICAL TRIAL: NCT01508481
Title: Vitamin D Inadequacy is Associated With Incidence of Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Principal Investigator, Seoul National University Bundang Hospital
Other Study IDs: VitaminD_T2DM
Record Dates: First submitted 2012-01-05; First posted 2012-01-12 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes
Keywords: Vitamin D; Diabetes; pancreas beta cell function; insulin resistance; Deficiency of Vitamin D3
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood sample was collected at the baseline.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes high risk group

SUMMARY:
Emerging evidence suggests that vitamin D [25-hydroxyvitamin D; 25(OH)D] may play a role in the etiology of type 2 diabetes. Vitamin D levels are lower in those with type 2 diabetes and impaired glucose tolerance (IGT) compared with those with normal glucose tolerance (NGT). In addition, a few prospective studies have shown a significant inverse association of baseline serum 25(OH)D with incident diabetes. To date, however, the exact mechanisms through which vitamin D affects diabetes risk are not yet fully known, particularly whether vitamin D plays a role in insulin resistance (IR) and/or b-cell dysfunction, the main pathophysiological disorders underlying type 2 diabetes. So, the investigators plan to examine the prospective associations of baseline vitamin D [25-hydroxyvitamin D; 25(OH)D] with insulin resistance (IR), b-cell function, and glucose homeostasis in subjects at risk for type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* one or more risk factors for diabetes, including:

  * obesity
  * hypertension
  * dislipidemia
  * a family history of diabetes

Exclusion Criteria:

* previous diagnosed diabetes
* vitamin D supplement.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants, aged over 30 years, are recruited from Korea, between January 2006 and December 2011. Participants are at high risk for type 2 diabetes, as they are recruited on the basis of the presence of one or more risk factors for diabetes, including obesity, hypertension, dislipidemia, and a family history of diabetes. Participants are contacted every 6 month after the baseline visit to update contact information and collect data on major health events. Participants are invited to return to the clinic examination centers after 3 years for follow-up assessments.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2007-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of diabetes | 5 years
  Incidence of diabetes defined by American Diabetes Association criteria

SECONDARY OUTCOMES:
Pancreatic beta cell function | 5 years
  Pancreatic beta cell function assessed by homeostasis model
Insulin resistance | 5 years
  Insulin resistance assessed by homeostasis model

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PHD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Lim S, Kim MJ, Choi SH, Shin CS, Park KS, Jang HC, Billings LK, Meigs JB. Association of vitamin D deficiency with incidence of type 2 diabetes in high-risk Asian subjects. Am J Clin Nutr. 2013 Mar;97(3):524-30. doi: 10.3945/ajcn.112.048496. Epub 2013 Jan 30. PMID 23364011